CLINICAL TRIAL: NCT00333125
Title: A Study of Glaucoma Therapy to Treat Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-25
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-05

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Travoprost; Timolol; Ophthalmic Solutions; Solutions; Duotrav; dorzolamide; dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Travoprost/Timolol (Experimental)
  Interventions: Drug: Travoprost 40 mcg/ml + Timolol 5 mg/ml eye drops, solution (DuoTrav); Other: Timolol Vehicle
- Dorzolamide/Timolol (Active Comparator)
  Interventions: Drug: Dorzolamide 20 mg/ml + Timolol 5 mg/ml eye drops, solution (Cosopt)

INTERVENTIONS:
Drug: Travoprost 40 mcg/ml + Timolol 5 mg/ml eye drops, solution (DuoTrav) — One drop in the study eye(s) once daily, 9 PM, for 6 weeks
  Other Names: DuoTrav
  Arms: Travoprost/Timolol
Drug: Dorzolamide 20 mg/ml + Timolol 5 mg/ml eye drops, solution (Cosopt) — One drop in the study eye(s) twice daily for 6 weeks
  Other Names: Cosopt
  Arms: Dorzolamide/Timolol
Other: Timolol Vehicle — One drop in the study eye(s) once daily for 6 weeks
  Arms: Travoprost/Timolol

SUMMARY:
The purpose of this study is to compare the intraocular pressure (IOP)-lowering efficacy and safety of two combination products in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older.
* Diagnosis of glaucoma or ocular hypertension.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Under 18.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2006-04; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Mean Intra-Ocular Pressure (IOP) | 6 weeks

REFERENCES:
- [Result] Saeed M, Kadir S, Kaufman SL, Murray RR, Milligan F, Cotton PB. Bleeding following endoscopic sphincterotomy: angiographic management by transcatheter embolization. Gastrointest Endosc. 1989 Jul-Aug;35(4):300-3. doi: 10.1016/s0016-5107(89)72796-6. PMID 2788589